CLINICAL TRIAL: NCT06838702
Title: Structured Data Collection of Patients Undergoing Liver Transplantation and Evaluated for Bone Mineral Metabolism
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: AEPOFE
Record Dates: First submitted 2024-12-03; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-11

CONDITIONS: Osteoporosis; Liver Transplant
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Observational cohort study offered consecutively to every liver transplant patient who arrives for the first endocrinology visit or returns for follow-up visit for bone metabolism assessment.

DETAILED DESCRIPTION:
The retrospective and prospective single-center observational cohort study will be offered consecutively to every liver transplant patient who arrives for the first endocrinology visit or returns for follow-up visit for bone metabolism assessment at UO Endocrinology of Policlinico S. Orsola-Malpighi.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients undergoing liver transplantation for any cause.
* Performance of bone densitometry
* Performance of examinations pertaining to mineral metabolism
* Obtaining informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver transplantation and followed at the Endocrinology Operating Unit for bone mineral metabolism.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2028-01-10 (Estimated); Study Completion 2028-01-11 (Estimated)

PRIMARY OUTCOMES:
Bone Mass in Liver Transplant Patients | through study completion, an average of 4 years
  Evaluation of bone mass in patients undergoing liver transplantation followed at the Endocrinology Operating Unit for Bone Mineral Metabolism, through the creation of a structured data collection in which to census all cases diagnosed and evaluated since 1/1/2009 at the U.O. Endocrinology of the S. Orsola-Malpighi Polyclinic. For the prospective phase, the expected duration of individual patient observation is 5 years
Calcium Metabolism Indices in Liver Transplant Patients | through study completion, an average of 4 years
  Evaluation of laboratory values related to calcium metabolism in patients undergoing liver transplantation, specifically focusing on blood levels of calcium, phosphate, parathyroid hormone (PTH), and vitamin D. These parameters will be assessed using standard laboratory tests conducted at the Endocrinology Operating Unit for Bone Mineral Metabolism. Data will be collected through a structured registry that includes all cases diagnosed and evaluated since 1/1/2009 at the U.O. Endocrinology of the S. Orsola-Malpighi Polyclinic.
Fracture Incidence in Liver Transplant Patients | through study completion, an average of 4 years
  Evaluation of fracture incidence in patients undergoing liver transplantation in patients undergoing liver transplantation followed at the Endocrinology Operating Unit for Bone Mineral Metabolism, through the creation of a structured data collection in which to census all cases diagnosed and evaluated since 1/1/2009 at the U.O. Endocrinology of the S. Orsola-Malpighi Polyclinic. For the prospective phase, the expected duration of individual patient observation is 5 years

SECONDARY OUTCOMES:
Prevalence of Fractures in Patients Undergoing Liver Transplantation | through study completion, an average of 4 years
  This measure will assess the correlation between liver transplantation and the prevalence of fractures in patients followed at the Endocrinology Unit. Fractures will be identified through clinical records and radiological assessments. The prevalence will be reported as the percentage of patients with fractures (%) within the study population.
Relationship Between Biochemical Parameters and Bone Mineral Density (BMD) Trends in Liver Transplant Patients | through study completion, an average of 4 years
  This measure will evaluate the correlation between specific biochemical parameters (e.g., calcium concentration in mg/dL, phosphate concentration in mg/dL, parathyroid hormone levels in pg/mL) and trends in bone mineral density (BMD) values in liver transplant patients. Bone Mineral Density (BMD) will be assessed using dual-energy X-ray absorptiometry (DEXA) scans, reported in g/cm². Biochemical parameters will be measured through blood tests, with each parameter reported in its respective unit of measure, with distinct units of measure and measurement tools explicitly identified.

CONTACTS AND LOCATIONS:
Overall Officials: Uberto Pagotto, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy